CLINICAL TRIAL: NCT02281097
Title: Transdermal Vagal Stimulation for the Treatment of Postural Tachycardia Syndrome
Brief Title: Transdermal Vagal Stimulation for POTS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Andre' Diedrich, Research Professor of Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: VANDERBILT_IRB_121816
Record Dates: First submitted 2014-10-21; First posted 2014-11-03 (Estimated); Last update posted 2025-02-05 (Actual); Status verified 2025-02

CONDITIONS: Postural Orthostatic Tachycardia Syndrome
Keywords: Postural Orthostatic Tachycardia Syndrome; POTS; Vagal Stimulation
MeSH Terms: conditions — Postural Orthostatic Tachycardia Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vagal Stimulation First (Active Comparator): Vagal stimulation to improve upright heart rate modulation and symptoms is given on first tilt study day.
  Placebo stimulation with ineffective low amplitude and frequency (sham intervention) is given on second tilt study.
  Interventions: Other: Stimulation; Other: Placebo
- Placebo First (Placebo Comparator): Placebo stimulation with ineffective low amplitude and frequency (sham intervention) is given on first tilt study day.
  Vagal stimulation to improve upright heart rate modulation and symptoms is given on second tilt study day.
  Interventions: Other: Stimulation; Other: Placebo

INTERVENTIONS:
Other: Stimulation — Application of current to skin above auricular branch of vagal nerve to modulate heart rate and symptoms
Other: Placebo — Application of low intensive current or frequency to skin above auricular branch of vagal nerve as sham intervention

SUMMARY:
Some patients experience high heart rates and symptoms of light-headedness, fatigue, headache during standing despite well maintained blood pressure.

These patient are disabled and can't be in upright position for a longer time. The purpose of this study is to test whether electrical stimulation of a nerve through a skin of the ear may improve heart rate response and reduce disabling symptoms.

DETAILED DESCRIPTION:
Background Postural Tachycardia Syndrome (POTS) is a syndrome characterized by disabling symptoms of inadequate cerebral perfusion on assuming the upright posture, including light-headedness, fatigue, palpitations, altered mentation, headache, nausea, presyncope, and occasionally syncope.

POTS is characterized by an excessive increase in heart rate and exaggerated increase in plasma catecholamine levels on standing in the absence of a blood pressure fall. These disabling symptoms persist for more than six months.

Objective The objective of this study is to study the effect of vagal stimulation on heart rate modulation during supine and upright posture as a treatment modality for patients with POTS.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking patients who qualify with the criteria of idiopathic postural tachycardia syndrome will be studied. The criteria are:

  1. an increase of heart rate of 30 beats/minute or an upright heart rate of >= 120 bpm, and
  2. chronic problems of symptoms during upright posture for at least 6 month.
* Subjects must also be able to safely withdrawn from medications that influence heart rate, blood pressure, and hormone levels that regulate blood pressure.
* The age limit is 18-75 years.

Exclusion Criteria:

* Patients that have other major medical problems, such as cancer or heart disease are excluded because the influence of that diagnosis on the symptoms is not known.
* Pregnancy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart Rate (average of 1 minute) | [-5,0,5,10,15,20,..,50 min] relative time from tilt
  Upright heart rate and heart rate change from supine measured during graded tilt with 15 degrees increments each 5 minutes till 30 min of 75 degrees or abort.

SECONDARY OUTCOMES:
Orthostatic Symptoms (Subjective analog symptoms scale (0-100) | [-5,0,5,10,15,20,..,50 min] relative time from tilt
  Subjective analog symptoms scale (0-100)
Orthostatic Tolerance (Maximal tolerated time in upright position) | [0-50 min] relative time from tilt
  Maximal tolerated time in upright position

CONTACTS AND LOCATIONS:
Overall Officials: Andre Diedrich, MD, PhD, Principal Investigator — Vanderbilt University Medical Center; Italo Biaggioni, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Autonomic Dysfunction Center, Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: No
No. There is no plan to share data.

REFERENCES:
- See also: Vanderbilt Autonomic Dysfunction Center — https://www.vumc.org/autonomic-dysfunction-center/vanderbilt-autonomic-dysfunction